CLINICAL TRIAL: NCT05912686
Title: High Dose of Atorvastatin for Preventing Cerebral Vascular Wall Damage in Patients Undergoing Mechanical Thrombectomy
Brief Title: High-Dose Atorvastatin for Vascular Wall Protection in Thrombectomy Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Dean, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PVD-MT
Record Dates: First submitted 2023-06-11; First posted 2023-06-22 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Mechanical Thrombectomy; Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Atorvastatin

STUDY DESIGN:
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-dose arm (Active Comparator): The test group will undergo high-dose atorvastatin treatment (80mg/day) for the first 3 days after the mechanical embolectomy, transitioning to a standard dose (20mg/day) of atorvastatin thereafter.
  Interventions: Drug: Atorvastatin 80mg
- standard-dose arm (Other): a standard dose (20mg/day) of atorvastatin after the mechanical embolectomy
  Interventions: Drug: Atorvastatin 20mg

INTERVENTIONS:
Drug: Atorvastatin 80mg — The test group will undergo high-dose atorvastatin treatment (80mg/day) for the first 3 days after the procedure, transitioning to a standard dose (20mg/day) of atorvastatin thereafter.
  Arms: high-dose arm
Drug: Atorvastatin 20mg — The control group will receive a consistent standard dose (20mg/day) of atorvastatin.
  Arms: standard-dose arm

SUMMARY:
This project investigates the impact of statins on cerebral vascular wall damage after mechanical thrombectomy. The investigators will undertake a multi-center, prospective, parallel-controlled, open-label, superiority randomized controlled study based on past research on intense lipid-lowering intervention trials. Patients undergoing post-thrombectomy will be divided into two groups: the test group and the control group. After surgery, the test group will be given a high dose of atorvastatin (80mg/day), followed by a standard dose (20mg/day). The control group will continue to receive the standard dose of atorvastatin (20mg/day). The investigators will compare the high-resolution vascular wall MRI characteristics (vascular wall enhancement, lumen stenosis rate, and so on) within 3-5 days of the operation, as well as the composite incidence of ischemic stroke, transient ischemic attack, intracranial hemorrhage 1 month postoperatively, and the modified Rankin Score at 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of acute ischemic stroke;
2. With anterior circulation acute stroke who meet and receive emergency endovascular treatment;
3. CTA or DSA confirms anterior circulation intracranial arterial lesions, including MT of intracranial arteries (middle cerebral artery (MCA), internal carotid artery (ICA), basilar artery and/or vertebral artery and P1 segment of posterior cerebral artery (PCA);
4. Recanalization of blood vessels after operation (mTICI ≥ 2b grade)

Exclusion Criteria:

1. Placing permanent stents or other implants in the target artery
2. Can not receive HR-VWI examination of 3T MRI due to claustrophobia or unstable condition
3. Contraindications to MRI and/or intravenous gadolinium

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Cerebral vascular wall damage | within 5-7 days after MT
  Incidence of T1 hyperintensity and T1 shortening within the arterial wall in HR-VWI

SECONDARY OUTCOMES:
Target vessel stenosis rate | Within 5-7 days after MT
  The stenosis rate of target blood vessel artery 5-7 days after MT surgery.
Perioperative complications | Within 30 days after MT
  Cumulative incidence rate of symptomatic intracranial hemorrhage, TIA or ischemic stroke within 30 days after MT surgery.
Neurological function evaluation | Within 90 days after MT
  Proportion of patients with good prognosis 3 months after MT surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, M.D., Principal Investigator — Zhongda hospital, Southeast university, Nanjing, China; Hai-Peng Wang, M.D., Principal Investigator — Zhongda hospital, Southeast university, Nanjing, China
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abraham P, Scott Pannell J, Santiago-Dieppa DR, Cheung V, Steinberg J, Wali A, Gupta M, Rennert RC, Lee RR, Khalessi AA. Vessel wall signal enhancement on 3-T MRI in acute stroke patients after stent retriever thrombectomy. Neurosurg Focus. 2017 Apr;42(4):E20. doi: 10.3171/2017.1.FOCUS16492. PMID 28366071
- [Background] Perren F, Kargiotis O, Pignat JM, Pereira VM. Hemodynamic Changes May Indicate Vessel Wall Injury After Stent Retrieval Thrombectomy for Acute Stroke. J Neuroimaging. 2018 Jul;28(4):412-415. doi: 10.1111/jon.12513. Epub 2018 Apr 14. PMID 29655219
- [Background] Krishnan R, Mays W, Elijovich L. Complications of Mechanical Thrombectomy in Acute Ischemic Stroke. Neurology. 2021 Nov 16;97(20 Suppl 2):S115-S125. doi: 10.1212/WNL.0000000000012803. PMID 34785610
- [Background] Lindenholz A, van der Schaaf IC, van der Kolk AG, van der Worp HB, Harteveld AA, Kappelle LJ, Hendrikse J. MRI Vessel Wall Imaging after Intra-Arterial Treatment for Acute Ischemic Stroke. AJNR Am J Neuroradiol. 2020 Apr;41(4):624-631. doi: 10.3174/ajnr.A6460. Epub 2020 Mar 5. PMID 32139427